CLINICAL TRIAL: NCT00412620
Title: Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of ABT-925 in Subjects With Acute Exacerbation of Schizophrenia
Brief Title: An Evaluation of the Safety and Efficacy of ABT-925 in Subjects With Acute Exacerbation of Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beatrice Rendenbach-Mueller, PhD, Project Director, Neuroscience/Anesthesia Department, Abbott Laboratories
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M06-816
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2010-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ABT-925

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo
- Group 1 Part 1 - ABT-925 (Experimental)
  Interventions: Drug: ABT-925
- Group 1 Part 2 - ABT-925 (Experimental)
  Interventions: Drug: ABT-925
- Group 2 - ABT-925 (Experimental)
  Interventions: Drug: ABT-925

INTERVENTIONS:
Drug: ABT-925
  Arms: Group 1 Part 1 - ABT-925; Group 1 Part 2 - ABT-925; Group 2 - ABT-925
Drug: Placebo
  Arms: Sugar Pill

SUMMARY:
The objective of this study is to explore the safety and efficacy of ABT-925 involving patients who meet the DSM-IV-TR (Diagnostic and Statistical Manual of Medical Disorders, Fourth Edition Text Revision) criteria for an acute exacerbation of schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
To explore the safety and efficacy of ABT-925 treatment at three different doses for 6 weeks compared with placebo in subjects with a diagnosis of acute exacerbation of schizophrenia or schizoaffective disorder according to DSM-IV-TR criteria (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision).

ELIGIBILITY:
Inclusion Criteria:

* The subject has a current primary diagnosis of schizophrenia or schizoaffective disorder; specifically, an acute exacerbation with prominent "active phase" symptoms, as described in Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision criteria (and confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision). Subjects with schizophrenia may belong to any of the following subtypes: paranoid, disorganized, catatonic, or undifferentiated.
* The subject has a The Positive and Negative Syndrome Scale total score of greater than or equal to 60.
* The subject has a score of greater than 4 ("moderate") on at least 2 out of the following 5 The Positive and Negative Syndrome Scale positive symptoms: delusions, conceptual disorganization, hallucinatory behavior, grandiosity, suspiciousness/persecution.
* The subject is between 18 and 65 years old inclusive at the time of randomization.
* The subject has a reliable caregiver (if applicable) or an identified responsible (e.g., family member, social worker, nurse) who will support him/her to ensure compliance with treatment and outpatient visits. In addition, the subject must have an adequate place of residence.
* The subject agrees to be hospitalized for the duration of the Taper off/Washout Period and at least the first fourteen days of the Double-blind Period.

Exclusion Criteria:

* The subject has a body mass index greater than 35.
* The subject has any condition that in the opinion of the investigator is likely to place him/her at an unacceptable safety risk by entering the study or by treatment with ABT-925.
* The subject has a diagnosis of one or more of the following conditions: another primary Axis I disorder, including schizophreniform disorder, bipolar disorder or major depressive disorder; comorbid Axis II diagnoses, including borderline personality disorder and mental retardation. (Note: a diagnosis of depression not otherwise specified is acceptable for inclusion into the study).
* The subject has a diagnosis of substance or alcohol disorder (abuse/dependence according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision criteria), excluding nicotine, within one (1) month prior to the beginning of the Screening Period, or in the opinion of the investigator, a disorder that will interfere with the conduct of the study.
* The subject has a history of substance-induced psychotic disorder in the previous 6 months.
* The subject has evidence suggestive of treatment-resistant schizophrenia (i.e., lack of significant clinical improvement despite adequate courses and doses of at least two different antipsychotic medications during the previous 2 years; or adequate use of clozapine indicated for treatment-resistant schizophrenia).
* The subject has serious violent, homicidal or suicidal ideation in the opinion of the investigator.
* The subject has a screening QT interval corrected by Bazett formula interval of greater than 430 msec if male and greater than 450 msec if female.
* The subject's Liver Function Tests (Aspartate aminotransferases, Alanine aminotransferase or total bilirubin levels) are not within normal limits at screening.
* The subject has a diagnosis, history, or a positive serological result suggestive of liver disease including but not limited to hepatitis and Gilbert's Syndrome.
* The subject has received any of the following treatments within the time periods described: mood stabilizers or antidepressants during the 30 days prior to Screening; electroconvulsive therapy during the 3 months prior to Screening; clozapine during 60 days prior to Screening.
* The subject is currently receiving treatment with oral psychotropic medications or has received depot neuroleptics within one inter-injection interval.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale | Assessed at screening and weekly from baseline through week 42/premature discontinuation
  The PANSS (The Positive and Negative Syndrome Scale) assesses the severity of symptoms of schizophrenia over the preceding seven days. The PANSS items are divided into positive, negative, and general psychopathology factors. The PANSS total score is the score of all 30 PANSS items taken together.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale | Assessed at screening and weekly from baseline through week 42/premature discontinuation
  Subscale of PANSS (The Positive and Negative Syndrome Scale)
Clinical Global Impression Severity score | Assessed at screening and weekly from baseline through week 42/premature discontinuation
  Assesses the overall, absolute degree of illness at any point in time (refer to the degree of illness at the time of the visit and during the week prior to the visit).
Calgary Depression Scale for Schizophrenia Total score | Assessed at screening and weekly from baseline through week 42/premature discontinuation
  The CDSS (Calgary Depression Scale for Schizophrenia Total score) consists of items designed to assess the severity of symptoms of depression in the presence of schizophrenia such as depressed mood, hopelessness, guilt, and insomnia.
Negative Symptom Assessment | Assessed at screening and weekly from baseline through week 42/premature discontinuation
  The NSA (Negative Symptom Assessment) is a 16-item instrument plus a one-item global rating designed to measure specific negative symptoms in schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Rendenbach-Mueller, PhD, Study Director — Abbott
Locations (18):
- United States (11):
  - Site Reference ID/Investigator# 5188, Anaheim, California
  - Site Reference ID/Investigator# 4539, Cerritos, California
  - Site Reference ID/Investigator# 4175, Garden Grove, California
  - Site Reference ID/Investigator# 4553, Pico Rivera, California
  - Site Reference ID/Investigator# 4173, San Diego, California
  - Site Reference ID/Investigator# 4565, Upland, California
  - Site Reference ID/Investigator# 4177, North Miami, Florida
  - Site Reference ID/Investigator# 4168, Atlanta, Georgia
  - Site Reference ID/Investigator# 4567, Austin, Texas
  - Site Reference ID/Investigator# 4176, Austin, Texas
  - Site Reference ID/Investigator# 4371, Bellaire, Texas
- Argentina (3):
  - Site Reference ID/Investigator# 5227, Buenos Aires
  - Site Reference ID/Investigator# 5226, Córdoba
  - Site Reference ID/Investigator# 5224, La Plata
- Mexico (4):
  - Site Reference ID/Investigator# 4305, Guadalajara
  - Site Reference ID/Investigator# 4304, Mexico City
  - Site Reference ID/Investigator# 4303, Mexico City
  - Site Reference ID/Investigator# 4298, Monterrey

REFERENCES:
- [Derived] Redden L, Rendenbach-Mueller B, Abi-Saab WM, Katz DA, Goenjian A, Robieson WZ, Wang Y, Goss SL, Greco N 4th, Saltarelli MD. A double-blind, randomized, placebo-controlled study of the dopamine D(3) receptor antagonist ABT-925 in patients with acute schizophrenia. J Clin Psychopharmacol. 2011 Apr;31(2):221-5. doi: 10.1097/JCP.0b013e31820e4818. PMID 21346607